CLINICAL TRIAL: NCT07352605
Title: Percutaneous Drainage Versus Antibiotic Therapy for Acute Diverticulitis With Abscess. The PANDA Randomized Controlled Trial Pilot Study
Brief Title: Percutaneous Drainage Versus Antibiotic Therapy for Acute Diverticulitis With Abscess.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Sanitaria di Firenze (Other)
Responsible Party: Principal Investigator, Alessio Giordano, Professor, Azienda Sanitaria di Firenze
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ASFirenze26
Record Dates: First submitted 2026-01-12; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Diverticular Disease of Colon
Keywords: Diverticulitis, Colonic diverticular abscess
MeSH Terms: conditions — Diverticulosis, Colonic; Diverticulitis | interventions — High-Energy Shock Waves; Random Allocation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Percutaneous drainage plus antibiotics. (Sham Comparator): Patients with diverticular abscess greater than 4 cm in diameter who undergo percutaneous drainage and antibiotic therapy
  Interventions: Procedure: Arm 1 (Control Arm) - Percutaneous drainage plus antibiotics: Image-guided (CT or ultrasound) percutaneous drainage performed within 48 hours of randomization with intravenous bro
- Antibiotics alone (Experimental): Patients with diverticular abscess larger than 4 cm in diameter who are undergoing antibiotic therapy alone
  Interventions: Other: Arm 2 (Experimental Arm) - Antibiotics alone: Intravenous broad-spectrum antibiotics: piperacillin-tazobactam 4 g/0.5 g q6h (dosage to be adjusted based on renal function) according to the recent lite

INTERVENTIONS:
Procedure: Arm 1 (Control Arm) - Percutaneous drainage plus antibiotics: Image-guided (CT or ultrasound) percutaneous drainage performed within 48 hours of randomization with intravenous bro — CT or ultrasound-guided percutaneous drainage
  Arms: Percutaneous drainage plus antibiotics.
Other: Arm 2 (Experimental Arm) - Antibiotics alone: Intravenous broad-spectrum antibiotics: piperacillin-tazobactam 4 g/0.5 g q6h (dosage to be adjusted based on renal function) according to the recent lite — Antibiotic therapy alone
  Arms: Antibiotics alone

SUMMARY:
the management of diverticular abscesses is guided by consensus-based recommendations from the WSES guidelines, the American College of Physicians, and the American Gastroenterological Association, all of which acknowledge the predominance of anecdotal and observational evidence and the urgent need for randomized controlled trials to inform clinical practice.The PANDA trial (Percutaneous drainage versus Antibiotic therapy for acute Diverticulitis with Abscess. Randomized controlled trial) is designed to address this evidence gap by directly comparing percutaneous drainage plus antibiotics versus antibiotics alone in patients with acute diverticulitis and large abscesses (WSES stage 2A). By employing strict inclusion criteria, standardized interventions, and predefined outcome measures, this study aims to clarify the relative efficacy, safety, and long-term impact of the two strategies, thereby guiding future clinical decision-making and informing guideline recommendations.

However, before we can proceed with the launch of the PANDA trial, we need to start a pilot study that will allow us to understand both the methodological and practical feasibility of starting this pilot study.

Primary objective The PANDA trial pilot study want to evaluate the local feasibility of the individual centers under study. Specifically, the primary objective will be to assess a minimum adherence rate of 70% for each participating center out of all patients with acute diverticulitis WSES 2A being evaluated. Adherence refers to the ability to enroll patients, randomize them, and perform clinical follow-up.

Secondary objectives The Panda trial pilot study want to compare the efficacy of antibiotic therapy alone versus percutaneous drainage plus antibiotic therapy in achieving complete clinical resolution at 30 days in patients with acute diverticulitis classified as WSES stage 2A, presenting with a pericolic or distant abscess ≥4 cm and < 8 cm in size.

In addition the PANDA trial pilot study wants to compare the rate of treatment failure, defined as the need for urgent surgical intervention (e.g., colectomy, resection with or without stoma formation) within 30 days.

Moreover the PANDA trial aimed to asses: the recurrence rate of diverticulitis after 90 days, defined as a new clinical episode confirmed radiologically and requiring hospital admission; to evaluate the length of hospital stay; to record and compare adverse events related to each treatment strategy, graded according to the Clavien-Dindo classification, with a focus on procedure-specific complications in the drainage arm.

Study Design

The PANDA trial pilot study is a prospective, multicentre, open-label, randomized controlled trial designed to compare two accepted non operative strategies for the management of large diverticular abscesses (WSES 2A Stage) to evaluate the methodological and structural feasibility of a national RCT. Participating centres will include high-volume emergency and general surgery units with access to both advanced interventional radiology and standardized medical management protocols. Two Intervention arms:

* Arm 1 (Control Arm) - Percutaneous drainage plus antibiotics.
* Arm 2 (Experimental Arm) - Antibiotics alone

In both arms the patients will be evaluated daily clinically and through laboratory tests.

Collaborators at each participating center will prospectively collect data for all eligible patients for 6 months followed by 3 months of follow-up.

ELIGIBILITY:
Inclusion criteria

* Patients of both sexes, ≥ 18 years old.
* Patients with abdominal CT scan diagnosis of colonic AD classifiable as WSES 2A with abscess ≥4 cm and < 8 cm in size;
* Patients with haemodynamic stability at hospital admission and no clinical or radiological evidence of diffuse peritonitis.
* Patients who accept and sign the informed consent

Exclusion criteria

* Patients with a final diagnosis other than diverticular abscess, including those diagnosed with colonic cancer.
* Pregnancy or lactation.
* Immunosuppressed patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-04 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Primary outcome | From enrollment to the end of treatment at 6 months
  The PANDA trial pilot study want to evaluate the local feasibility of the individual centers under study. Specifically, the primary objective will be to assess a minimum adherence rate of 70% for each participating center out of all patients with acute diverticulitis WSES 2A being evaluated. Adherence refers to the ability to enroll patients, randomize them, and perform clinical follow-up.

SECONDARY OUTCOMES:
Secondary outcomes | From enrollment to the end of treatment at 9 months
  The Panda trial pilot study want to compare the efficacy of antibiotic therapy alone versus percutaneous drainage plus antibiotic therapy in achieving complete clinical resolution at 30 days in patients with acute diverticulitis classified as WSES stage 2A, presenting with a pericolic or distant abscess ≥4 cm and < 8 cm in size.
  In addition the PANDA trial pilot study wants to compare the rate of treatment failure, defined as the need for urgent surgical intervention (e.g., colectomy, resection with or without stoma formation) within 30 days.
  Moreover the PANDA trial aimed to asses: the recurrence rate of diverticulitis after 90 days, defined as a new clinical episode confirmed radiologically and requiring hospital admission; to evaluate the length of hospital stay; to record and compare adverse events related to each treatment strategy, graded according to the Clavien-Dindo classification, with a focus on procedure-specific complications in the drainage arm.

IPD SHARING:
Plan to Share IPD: Undecided